CLINICAL TRIAL: NCT00458237
Title: A Brief Dose Escalation Followed by a Phase 2 Study of RAD001 in Combination With Trastuzumab in HER2-Positive Metastatic Breast Cancer
Brief Title: Dose Escalation Followed by Study of RAD001 in Combination With Trastuzumab in HER2-Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Gerburg Wulf, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-124
Record Dates: First submitted 2007-04-09; First posted 2007-04-10 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: HER2 positive; metastatic breast cancer; RAD001; Herceptin
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ph I: Everolimus L1 + Trastuzumab (Experimental): Cycle duration is 21 days. Participants receive trastuzumab 6 mg/kg [8 mg/kg loading dose] IV once every three weeks and take everolimus 5 mg by mouth daily on days 1-21. Participants are treated until disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus; Drug: Trastuzumab
- Ph I: Everolimus L2 + Trastuzumab (Experimental): Cycle duration is 21 days. Participants receive trastuzumab 6 mg/kg [8 mg/kg loading dose] IV once every three weeks and take everolimus 10 mg by mouth daily on days 1-21. Participants are treated until disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus; Drug: Trastuzumab
- PhII: Everolimus MTD + Trastuzumab (Experimental): Cycle duration is 21 days. Participants receive trastuzumab 6 mg/kg [8 mg/kg loading dose] IV once every three weeks and take everolimus at the MTD by mouth daily on days 1-21. Participants are treated until disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus; Drug: Trastuzumab

INTERVENTIONS:
Drug: Everolimus — Everolimus is being administered orally 7 days per week.
  Other Names: RAD001
Drug: Trastuzumab — Trastuzumab is being administered at a dose of 6 mg/kg intravenously once every 21 days.
  Other Names: Herceptin

SUMMARY:
The purpose of this research study is to determine the safety of RAD001 and the highest dose of this drug that can be given to people with HER2-positive metastatic breast cancer safely in combination with trastuzumab. RAD001 has been used in patients with severe rheumatoid arthritis, in recipients of solid-organ transplants, healthy volunteers and experiments with animals, and information from those other research studies suggest that this RAD001 may help to stop cancer cells from growing abnormally.

DETAILED DESCRIPTION:
* Since we are looking for the dose of RAD001 that can be given safely in combination with trastuzumab, not everyone will receive the same amount of RAD001. Small groups of participants will be enrolled at a certain dose of RAD001 and if they tolerate the medications well, the next small group will receive a higher dose. This will continue until the optimal dose of RAD001 that can be given in combination with trastuzumab is found.
* Blood will be drawn on days 1, 2, 8, and 15 of the first cycle of treatment and then once at every 4 cycles for everolimus pharmacokinetics analysis.
* There is an optional tissue biopsy component to this study asking for 2 biopsies performed pre-treatment and after the cycle one.
* We will keep track of the participants medical condition for the next three years by calling them on the telephone twice a year to see how they are doing.

OBJECTIVES:

Primary

- To assess the safety and tolerability of RAD001 in combination with trastuzumab in HER2-positive metastatic breast cancer

Secondary

* To evaluate the activity of RAD001 plus trastuzumab, as defined by objective response rate, in patients with progression on a trastuzumab-containing regimen
* To evaluate changes in signaling molecules in response to trastuzumab and RAD001 in circulating tumor cells and tumor tissue
* To evaluate the pharmacokinetics of RAD001 in combination with trastuzumab.

STATISTICAL DESIGN:

This Phase I study followed a standard 3+3 dose escalation design with two dose levels of everolimus in combination with trastuzumab to be evaluated. The DLT observation period was cycle one (first 21 days of treatment). There is a 20 patient expansion cohort treated at the MTD. The regimen would be considered promising if at least 2 objective responses are observed out of 20 treated patients. If the true but unknown response rate is 15% then the probability of observing at least 2 responses is 82% but if the true rate is 5% this probability reduces to 26%.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast cancer, with stage IV disease
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as greater than or equal to 20mm with conventional techniques or as greater than or equal to 10mm with spiral CT scan.
* Primary tumor or metastasis must overexpress HER2
* Patient must have received 1-2 prior chemotherapeutic regiments for metastatic breast cancer and must have been off treatment for at least three weeks.
* Patient must have received and progressed on at least 1 prior trastuzumab-containing regimen, but not more than 2, in the metastatic setting.
* Patients may have received prior radiation therapy
* Patients may have received hormonal therapy in the adjuvant or metastatic setting
* 18 years of age or older
* Life expectancy of greater than 6 months
* Normal organ and marrow function as defined in the protocol
* Left ventricular ejection fraction (LVEF) greater than or equal to the institutional lower limit of normal

Exclusion Criteria:

* Treatment with any investigational drug within 4 weeks
* Long-term treatment, over 3 months, with a systemic steroid or another immunosuppressive agent
* Other malignancies within the past 3 years, except for adequately treated carcinoma of teh cervix or basal-or squamous-cell carcinoma of the skin
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001
* An active, bleeding diathesis or an oral anti-vitamin K medication
* Prior treatment with an mTOR inhibitor
* History of non-compliance with medical regimens
* Unwillingness or inability to comply with the protocol
* Major surgery within 2 weeks before study entry
* Patients with active brain metastases or leptomeningeal carcinomatosis
* Patients who have experienced grade 1 or grade 2 hypersensitivity reactions to prior trastuzumab therapy are eligible ONLY IF these reactions did not prevent further administration
* Severe and/or uncontrolled intercurrent medical condition, psychiatric illness or a social situation that could limit their ability to comply with the study requirements.
* Pregnant or breast-feeding women
* HIV positive patients
* Known hypersensitivity to RAD001 (everolimus) or other rapamycins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerburg Wulf, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Morrow PK, Wulf GM, Ensor J, Booser DJ, Moore JA, Flores PR, Xiong Y, Zhang S, Krop IE, Winer EP, Kindelberger DW, Coviello J, Sahin AA, Nunez R, Hortobagyi GN, Yu D, Esteva FJ. Phase I/II study of trastuzumab in combination with everolimus (RAD001) in patients with HER2-overexpressing metastatic breast cancer who progressed on trastuzumab-based therapy. J Clin Oncol. 2011 Aug 10;29(23):3126-32. doi: 10.1200/JCO.2010.32.2321. Epub 2011 Jul 5. PMID 21730275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from July 2007 through May 2009.
Groups:
- Phase I: Everolimus (Dose Level 1) and Trastuzumab: Cycle duration is 21 days. Participants receive trastuzumab 6 mg/kg [8 mg/kg loading dose] IV once every three weeks and take everolimus 5 mg by mouth daily on days 1-21. Participants are treated until disease progression or unacceptable toxicity.
- Phase I: Everolimus (Dose Level 2) and Trastuzumab: Cycle duration is 21 days. Participants receive trastuzumab 6 mg/kg [8 mg/kg loading dose] IV once every three weeks and take everolimus 10 mg by mouth daily on days 1-21. Participants are treated until disease progression or unacceptable toxicity.
- Phase II: Everolimus (Maximum Tolerated Dose) and Trastuzumab: Cycle duration is 21 days. Participants receive trastuzumab 6 mg/kg [8 mg/kg loading dose] IV once every three weeks and take everolimus at the MTD (10 mg) by mouth daily on days 1-21. Participants are treated until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase I: Everolimus (Dose Level 1) and Trastuzumab | Phase I: Everolimus (Dose Level 2) and Trastuzumab | Phase II: Everolimus (Maximum Tolerated Dose) and Trastuzumab
Started | 3 | 3 | 5
Completed | 3 | 3 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Everolimus (Dose Level 1) and Trastuzumab | Phase I: Everolimus (Dose Level 2) and Trastuzumab | Phase II: Everolimus (Maximum Tolerated Dose) and Trastuzumab | Total
Number analyzed (Participants) | 3 | 3 | 5 | 11
Age, Continuous [Mean (Full Range); unit: years] | 53 [43 to 61] | 42 [40 to 43] | 42 [28 to 54] | 45 [28 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 11
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD is determined by the number of patients who experience a dose limiting toxicity (DLT). The MTD is defined as the highest dose at which fewer than one-third of patients experience a DLT. If no DLTs are observed, the MTD is not reached. Dose Limiting Toxicities (DLTs) were defined as follows (CTCAE v4.0):
  * Any grade 4 hematologic toxicity, excluding anemia.
  * Any grade 3 or 4 nonhematologic toxicity, except for nausea, vomiting, diarrhea, or hyperlipidemia that responds promptly (within 24 hours for nausea, vomiting, and diarrhea and within 1 week for hyperlipidemia) to appropriate treatment, and except for cardiac toxicity which will be assessed after 12 weeks of treatment.
  * Need to hold >1 dose of trastuzumab or > 7 doses of RAD001 within the first 3 weeks because of the presence of toxicity.
Time Frame: Cycle One (first 21 days of treatment)
Population: The analysis dataset for the Phase I study is comprised of the two dose cohorts: Level 1 and 2.
Measure: Number; unit: participants with DLT
Arm/Group | Phase I: Everolimus (Dose Level 1) and Trastuzumab | Phase I: Everolimus (Dose Level 2) and Trastuzumab
Number analyzed (Participants) | 3 | 3
participants with DLT | 0 | 0

2. Secondary Outcome: Clinical Response Rate
Description: Best response on treatment was based on RECIST 1.0 criteria with overall clinical response defined as achieving stable disease (SD), partial response (PR) or complete response (CR). Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response. SD is neither CR/PR or progressive disease (PD). PD is at least a 20% increase in sum LD, takings as reference smallest sum LD since treatment started.
Time Frame: Disease assessments occurred every 9 weeks (3 cycles) on treatment. Treatment continued until disease progression or unacceptable toxicity. Median duration of treatment was 2.4 months.
Population: The analysis dataset is comprised of patients treated at the MTD/dose level 2.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Phase I: Everolimus (Dose Level 2) and Trastuzumab | Phase II: Everolimus (Maximum Tolerated Dose) and Trastuzumab
Number analyzed (Participants) | 3 | 5
proportion of participants | .67 [.14 to .98] | .80 [.34 to .99]

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment. Median duration of treatment was 2.4 months.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3.
Arm/Group | Phase I: Everolimus (Dose Level 1) and Trastuzumab | Phase I: Everolimus (Dose Level 2) and Trastuzumab | Phase II: Everolimus (Maximum Tolerated Dose) and Trastuzumab
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 4/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Everolimus (Dose Level 1) and Trastuzumab (N=3) | Phase I: Everolimus (Dose Level 2) and Trastuzumab (N=3) | Phase II: Everolimus (Maximum Tolerated Dose) and Trastuzumab (N=5)
Fatigue (General disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Leukocytes (Investigations) | 0 | 0 | 1
Lymphopenia (Investigations) | 0 | 1 | 0
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 0 | 0 | 1
Neutrophils (Investigations) | 0 | 0 | 1
Platelets (Investigations) | 0 | 0 | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 0 | 2 — Note these are the same 2 cases of Vascular access, Thrombosis/embolism occurring on the same cycle but here grade 4.
Vascular access-Thrombosis/embolism (Injury, poisoning and procedural complications) | 0 | 0 | 2 — Note these are the same 2 cases of Thrombosis/thrombus/embolism occurring on the same cycle but here grade 3.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Everolimus (Dose Level 1) and Trastuzumab (N=3) | Phase I: Everolimus (Dose Level 2) and Trastuzumab (N=3) | Phase II: Everolimus (Maximum Tolerated Dose) and Trastuzumab (N=5)
ALT- SGPT (Investigations) | 0 | 1 | 3
AST- SGOT (Investigations) | 3 | 2 | 4
Abdomen- pain (Gastrointestinal disorders) | 0 | 1 | 0
Alkaline phosphatase (Investigations) | 0 | 1 | 1
Allergic reaction (Immune system disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bicarbonate (Metabolism and nutrition disorders) | 0 | 1 | 1
Breast- pain (Reproductive system and breast disorders) | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cardiac-other (Cardiac disorders) | 0 | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 0 | 1 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Edema head and neck (General disorders) | 0 | 0 | 1
Edema limb (General disorders) | 0 | 0 | 1
Extremity-limb- pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 2
Fever w/o neutropenia (General disorders) | 0 | 1 | 1
Gallbladder- pain (Hepatobiliary disorders) | 0 | 0 | 1
Head/headache (Nervous system disorders) | 0 | 2 | 0
Hematologic-other (Blood and lymphatic system disorders) | 0 | 1 | 1
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1 | 4
Hot flashes (Vascular disorders) | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolemia (Investigations) | 2 | 3 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Infection Gr0-2 neut- skin (Infections and infestations) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Leukocytes (Investigations) | 0 | 1 | 3
Liver- pain (Hepatobiliary disorders) | 0 | 0 | 1
Lymphedema-related fibrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lymphopenia (Investigations) | 1 | 0 | 0
Metabolic/Laboratory-other (Investigations) | 0 | 0 | 2
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 0 | 2 | 0
Muco/stomatitis by exam- oral cavity (Gastrointestinal disorders) | 0 | 0 | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Neuropathy-sensory (Nervous system disorders) | 0 | 0 | 1
Neutrophils (Investigations) | 1 | 1 | 0
Pain NOS (General disorders) | 0 | 1 | 0
Platelets (Investigations) | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rectum- pain (Gastrointestinal disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Skin-other (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Taste Disturbance (Nervous system disorders) | 1 | 0 | 0
Throat/pharynx/larynx- pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 1 | 0
Vaginal discharge (non-infectious (Reproductive system and breast disorders) | 0 | 1 | 0
Vision-photophobia (Eye disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Weight loss (Investigations) | 0 | 0 | 1
Pain-Larynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pain-Joint (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No